CLINICAL TRIAL: NCT03943992
Title: A Randomized, Double-blind, Double-dummy, Active Comparator, Multi-centers, Non-inferiority Design Clinical Trial to Assess the Efficacy and Safety of YYD601 in the Treatment of Esophageal Reflux Disease (ERD) (Phase3).
Brief Title: Clinical Trial to Assess the Efficacy and Safety of YYD601 in the Treatment of Esophageal Reflux Disease (ERD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yooyoung Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YYPCT_YYD601_P3
Record Dates: First submitted 2019-03-25; First posted 2019-05-09 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Erosive Esophagitis
MeSH Terms: interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- YYD601 40mg (Experimental): Esomeprazole magnesium Dihydrate.
  Interventions: Drug: YYD601 40mg; Drug: Placebos
- Nexium 40mg (Active Comparator): Esomeprazole magnesium trihydrate, a substituted benzimidazole.
  Interventions: Drug: Nexium 40mg; Drug: Placebos

INTERVENTIONS:
Drug: YYD601 40mg — Patients should take druges 30 minutes before breakfast.
  Arms: YYD601 40mg
Drug: Nexium 40mg — Patients should take druges 30 minutes before breakfast.
  Arms: Nexium 40mg
Drug: Placebos — The placebo YYD601 is made from microcrystalline cellulose covered with hard shell. The placebo Nexium is made from microcrystalline cellulose, Crospovidone, Magnesiumstearat and other ingredients.

SUMMARY:
A randomized, double-blind, double-dummy, active comparator, multi-centers, non-inferiority design clinical trial to assess the efficacy and safety of YYD601 in ERD patients (phase 3).

DETAILED DESCRIPTION:
This phase 3 clinical trial is designed as randomized, active-comparator, double-dummy, multi-center for ERD patients, who take YYD601 40mg or Nexium 40mg for 8 weeks. Each part is assessed by 'LA grade' measured through the endoscopy, target goal is to confirm the non-inferiority of YYD601 40mg to Nexium 40mg.

ELIGIBILITY:
Inclusion Criteria:

* A man or woman over 20 years old less than 70 years old.
* A man or woman who has experienced symptom (heartburn and acid regurgitation) within 7 days before Visit 1, meet below 1) or 2) criteria, who has been made diagnosis as Erosive esophagitis(LA grade A~D) measured through the endoscopy which is carried out within (-2W±D2)

  * Symptom (heartburn and acid regurgitation) is confirmed by RDQ.
  1. Experienced above 2 days in 1 week, Heartburn of acid regurgitation above the weakness.
  2. Experienced above 1 day in 1 week, Heartburn of acid regurgitation above the middle.
* A man or woman who has a full understanding of this clinical trial through the detailed explanation, agree in writing to participate in this trial.

Exclusion Criteria:

* Who has hyper sensitivity reaction about other drugs, ingredients, components of investigator product or compound of benzimidazole.
* Who has NERD
* Who get a diagnosis as a IBS within the last 3 months.
* Who have taken gastric acid secretion inhibitors including PPIs within 2 weeks before the endoscopy.
* Who have taken drugs about reflux esophagitis (H₂-receptor inhibitor (H2RA) Prostaglandin(PG), Antacid, Prokinetic acid etc.) above 2 times as an usual dose. (* refer to the Concomitant medication in text.)
* Who has been experienced the disease affecting the esophagus(Eosinophilic esophagitis, esophageal varices, cirrhosis, Virus or Fungal infection, Esophageal stricture, primary esophageal motility disorder and gastrointestinal bleeding). Or who has a history of radio therapeutics, freeze treatment about the esophagus.
* Who has clinically significant abnormal result of ECG.
* Abnormal result of Major arrhythmia, Multifocal PVS, 2 AV-blcok etc.
* Who has the Schatzki near the LES(lower esophageal sphincter) except the Barret's esophagus.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
LA grade 0(zero) | within 8 weeks
  Percentage of patients(%) who's erosive esophagitis has been recovered to LA grade 0(zero) within week 8.
  Calculation of the sample size was based on a margin of non-inferiority by Normal approximation.

SECONDARY OUTCOMES:
LA grade 0(zero) | at 4 weeks
  Percentage of patients(%) who's erosive esophagitis has been recovered to LA grade 0(zero) by Normal approximation and Fisher's exact test.
Frequency variation of the Heartburn and acid regurgitation by RDQ(questionnaire). | at week 4 and 8 from baseline
  Change in frequency of the symptom(heartburn and acid regurgitation) by Shapiro-Wilk test and Wilcoxon's rank sum test.
Frequency variation of the Heartburn in daytime by patients diary | at 4 week and 8 week from baseline
  Percentage of patients(%) who have the symptom(heartburn and acid regurgitation) by Chi-square test and Fisher's exact test.
Frequency variation of the Heartburn in nighttime by patients diary | at 4 week and 8 week from baseline
  Percentage of patients(%) who have the symptom(heartburn and acid regurgitation) by Chi-square test and Fisher's exact test.
Days percentage(%) of no symptoms about the Heartburn and acid regurgitation | at week 4 and 8 from baseline
  Patients who have experienced the heartburn and acid regurgitation in nighttime by patients diary.

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Ansan Hospital, Seoul, South Korea